CLINICAL TRIAL: NCT05585580
Title: Efficacy and Safety of Serplulimab, Lenvatinib, and Paclitaxel in the Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma After First-line Immunotherapy: a Prospective, Single-armed Clinical Trial
Brief Title: Second-line Treatment With Serplulimab, Lenvatinib, and Paclitaxel in Advanced Gastric Cancer After Prior Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STILL
Record Dates: First submitted 2022-09-06; First posted 2022-10-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — lenvatinib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab, lenvatinib and paclitaxel/Paclitaxel for Injection (Albumin Bound)/Paclitaxel liposome (Experimental): Patients will be treated with serplulimab combined with lenvatinib and paclitaxel/ Paclitaxel for Injection (Albumin Bound)/Paclitaxel liposomefor 6 cycles, followed by serplulimab combined with lenvatinib maintenance therapy until disease progression, intolerable adverse reactions, or withdrawal of treatment consent.
  Interventions: Drug: Serplulimab; Drug: Lenvatinib; Drug: Paclitaxel/Paclitaxel-albumin/Paclitaxel liposome

INTERVENTIONS:
Drug: Serplulimab — 300mg d1 q3w
Drug: Lenvatinib — 8mg po qd
Drug: Paclitaxel/Paclitaxel-albumin/Paclitaxel liposome — 135~175mg/m2 /260mg/m2/135-175mg/m2 d1 q3w

SUMMARY:
This is a prospective, single arm, multicenter phase II study to assess the effectiveness of Serplulimab, Lenvatinib and Paclitaxel in the treatment of advanced gastric or gastroesophageal junction adenocarcinoma after first-line immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, gender is not limited;
2. Histologically or cytologically proven metastatic or locally advanced gastric or gastroesophageal junction adenocarcinoma
3. Programmed death-ligand 1 (PD-L1) positive subjects (CPS ≥ 1), or those who have achieved objective response to first-line Programmed death-1 (PD-1)/PD-L1 inhibitor therapy， or previous first-line PD-1/PD-L1 inhibitor therapy Treatment of PFS ≥ 6 months;
4. Prior chemotherapy, surgery, radiotherapy, or immunotherapy-related toxicity (excluding alopecia) has resolved to CTCAE ≤ grade 1;
5. Has measurable disease as determined by RECIST 1.1；
6. Subjects who can provide tissue samples (preferably freshly obtained tumor tissue before second-line therapy) for central laboratory testing for PD-L1 expression level determination；
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
8. Adequate organ function:

   1. Blood routine (no blood transfusion within 14 days before treatment, no granulocyte colony-stimulating factor, no correction with other drugs) i. Neutrophil count (NE)>1.5*109/L; ii. Hemoglobin count (HGB) > 90 g/L; iii. Platelet count (PLT)>100*109/L;
   2. Coagulation function (no blood product transfusion within 14 days before treatment) i. International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5*Upper Limit of Normal (ULN);
   3. Blood biochemistry (liver and kidney function) i. Creatinine clearance ≥50 mL/min; ii. Total bilirubin (TBIL)≤1.5×ULN; iii. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP)≤2.5*ULN; iv. Albumin > 2.7 g/dL
9. The urine protein of the patient is less than or equal to 1+;
10. According to the judgment of the investigator, the life expectancy is ≥6 months;
11. Able and willing to give written informed consent and has signed the informed consent form (ICF), prior to performance of any trial activities.
12. Female patients must be surgically sterilized females, postmenopausal, or using some form of highly effective contraception during treatment and within 12 weeks after treatment; male patients must be surgically sterilized men, or during treatment and 6 months after treatment effective contraceptive method

Exclusion Criteria:

1. Human epidermal growth factor receptor 2 (HER2) positive;
2. History of treatment with multi-target small molecule inhibitors such as lenvatinib or paclitaxel drugs;
3. Received systemic therapy (including chemotherapy, immunotherapy or targeted therapy) or local therapy (including surgery, radiotherapy) for advanced disease within 14 days before enrollment;
4. Hypertension that is difficult to control by drugs (systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 90 mmHg);
5. Patients with brain metastases, cancerous meningitis, spinal cord compression, or diseases of the brain or leptomeninges found in imaging CT or MRI examinations during screening;
6. Associated with refractory pleural effusion or ascites, such as pleural effusion or ascites that requires puncture and drainage within 2 weeks before the first administration;
7. Have other malignancies except cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors (Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading basement membrane));
8. Allergy to any study drug or excipients;
9. Chronic hepatitis B or HBV carriers with chronic hepatitis B virus (HBV) DNA exceeding 500 IU/mL, or patients with active hepatitis C virus (HCV) infection;
10. Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, thyroid function Hyperthyroidism, hypothyroidism), or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or other investigators' assessment that they have an impact on the study treatment;
11. Long-term heavy use of hormones or use of other immunomodulators;
12. Active infection;
13. Have been vaccinated with live or attenuated vaccines within 30 days before the first dose, or plan to receive live or attenuated vaccines during the study period, excluding the new crown vaccine;
14. Arterial/venous thrombotic events within 6 months, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism;
15. Severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, or stent placement within 6 months before enrollment; poorly controlled arrhythmia; according to the New York Heart Association (NYHA) criteria, III to IV Grade 1 cardiac insufficiency, or echocardiography showed left ventricular ejection fraction (LVEF) <50%;
16. History of interstitial lung disease or uncontrolled systemic disease, including diabetes, acute lung disease, etc.;
17. Known human immunodeficiency virus (HIV) infection;
18. Any major surgery requiring general anesthesia has been performed within ≤ 28 days before the first dose;
19. There is an underlying medical condition or alcohol/drug abuse or dependence that is not conducive to the administration of the study drug, or may affect the interpretation of the results, or put the patient at a high risk of treatment complications;
20. Participated in other therapeutic clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate （ORR) | 6 months after the last subject participating in
  Objective response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months after the last subject participating in
  Progression-free survival
Overall survival (OS) | 24 months after the last subject participating in
  Overall survival
Disease Control Rate (DCR) | 6 months after the last subject participating in
  Disease Control Rate
Duration of Overall Response (DOR) | 6 months after the last subject participating in
  Duration of Overall Response
Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE | through study completion, an average of 1 year.
  Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Lian Liu, Principal Investigator — Qilu hospital of Shandong univertisy
Locations (7):
- China (7):
  - Qilu hospital of Shandong univertisy, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao Municipal Hospital（Group）, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Linyi Cancer Hospital, Linyi

IPD SHARING:
Plan to Share IPD: No